CLINICAL TRIAL: NCT03490461
Title: Effects of Statin on Hepatocellular Carcinoma Recurrence After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0942
Record Dates: First submitted 2018-03-29; First posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Statin group: Statin therapy was defined as the administration of statins for more than 30 days after liver transplantation
  Interventions: Drug: Statin
- Non-statin group: the administration of statins for less than 30 days after liver transplantation

INTERVENTIONS:
Drug: Statin — Patients who used statins over 1 month for the treatment of dyslipidemia after LT were enrolled as statin group.
  Groups: Statin group

SUMMARY:
This study aims to investigate whether statin therapy can help prevent recurrence of hepatocellular carcinoma (HCC) in transplant recipients who had liver transplantation for HCC. Multiple logistic regression analysis will be performed to evaluate the association between statin therapy and the risk of HCC recurrence after LT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received LT at the Severance Hospital from 2006 to 2016.

Exclusion Criteria:

* early postoperative mortality (defined as death within 2 months after LT without signs of tumor recurrence)
* patient with distant lymph node metastasis confirmed within 1 month after LT
* Patients younger than 20 years of age
* patients who had LT for cirrhosis without confirmed HCC

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received LT at the Severance Hospital from 2006 to 2016.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
A new lesion with radiographic features compatible with HCC was defined as recurrence of HCC. | up to December, 2017
  Usually, liver CT is performed at 1 week, 1 month, 6 months, and every year until 5 years after surgery. Afterwards, liver CT is performed at 2-year intervals. Measurement of blood tumor markers [AFP and prothrombin induced by vitamin K absence-II] is performed every month for 6 months after discharge from the hospital and every 3 months thereafter. Additional liver CT, liver magnetic resonance imaging, or positron emission tomography-CT is performed when elevated tumor markers or suspicious lesions were noted. A new lesion with radiographic features compatible with HCC is defined as recurrence of HCC based on the reports of specialist in radiology.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology and Metabolism Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No